CLINICAL TRIAL: NCT06622304
Title: Mendelian Randomization Analysis of Drug Targets: Exploring the Impact of Antihypertensive and Lipid-Lowering Therapies on Inflammatory Cytokines
Brief Title: Exploring the Effects of Antihypertensive and Lipid-Lowering Drugs on Inflammatory Cytokine Levels
Acronym: MRDLT
Status: Completed | Type: Observational
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Collaborators: Shanghai Guanghua Hospital of Integrated Traditional Chinese and Western Medicine (Other)
Responsible Party: Principal Investigator, Zhibin Xu, Professor, Guangzhou Institute of Respiratory Disease
Other Study IDs: YYKC-2021-01-102
Record Dates: First submitted 2024-09-29; First posted 2024-10-02 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Hypertension; Dyslipidemias; Inflammatory Response; Chronic Inflammation; Inflammatory Cytokines
Keywords: Antihypertensive Drugs; Lipid-Lowering Drugs; Mendelian Randomization; ACE Inhibitors; ARBs; HMG-CoA Reductase Inhibitors; PCSK9 Inhibitors; NPC1L1 Inhibitors; IL-1β; TNF-α; CRP; MCP-1; Inflammatory Pathways; Genetic Association Studies; Causal Inference
MeSH Terms: conditions — Hypertension; Dyslipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — No biospecimen retention. The study utilizes existing genome-wide association study (GWAS) and expression quantitative trait loci (eQTL) data, with no collection of new biological specimens.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study investigates the causal relationships between antihypertensive and lipid-lowering drugs and inflammatory cytokines using a drug-targeted Mendelian randomization approach. By leveraging genome-wide association studies (GWAS) and expression quantitative trait loci (eQTL) data, the study evaluates the effects of angiotensin-converting enzyme inhibitors (ACEIs), angiotensin receptor blockers (ARBs), HMG-CoA reductase inhibitors, PCSK9 inhibitors, and NPC1L1 inhibitors on key inflammatory cytokines such as IL-1β, TNF-α, CRP, and MCP-1. The findings aim to provide insights into the prevention and control of excessive inflammatory responses, particularly in patients with hypertension and dyslipidemia, by assessing the causal effects of these therapies.

DETAILED DESCRIPTION:
This observational study focuses on elucidating the causal relationships between commonly prescribed antihypertensive drugs (ACEIs and ARBs) and lipid-lowering drugs (HMG-CoA reductase inhibitors, PCSK9 inhibitors, and NPC1L1 inhibitors) with various inflammatory cytokines, including IL-1β, TNF-α, CRP, MCP-1, and IFN-γ, using a drug-targeted Mendelian randomization (MR) framework. The study employs large-scale genetic data from European populations, drawing from genome-wide association studies (GWAS) and expression quantitative trait loci (eQTL) datasets, to construct instrumental variables that mimic the effects of drug exposure.

The primary aim is to explore how these pharmaceutical interventions influence inflammatory pathways at the molecular level. The use of MR methods enables causal inference by utilizing genetic variants within or near drug-target genes, allowing for the estimation of downstream effects similar to those produced by actual drug interventions. Key statistical methods, including inverse variance weighting and sensitivity analyses, are applied to ensure robustness and validity of the results.

This research provides critical evidence for the selection of antihypertensive and lipid-lowering therapies that not only manage cardiovascular risk factors but also modulate inflammation, contributing to personalized medicine strategies for patients with chronic inflammatory conditions. Furthermore, the findings have broader implications for drug repurposing and the development of new therapeutic targets aimed at mitigating inflammatory processes that underlie various chronic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 years or older.
* Diagnosed with hypertension, coronary artery disease, or dyslipidemia.
* Availability of complete genome-wide data and inflammatory cytokine levels.
* Willingness to participate in the study and provide the required clinical data.

Exclusion Criteria:

* Participants under the age of 18.
* Individuals with severe chronic diseases or other conditions that may significantly influence inflammatory responses.
* Individuals unwilling or unable to provide necessary clinical or genomic data.
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adult patients diagnosed with hypertension, coronary artery disease, or dyslipidemia. These participants have genome-wide data collected through genome-wide association studies (GWAS) and include measurements of inflammatory cytokines. The study focuses on the effect of drug interventions on inflammatory biomarkers.
Sampling Method: Non-Probability Sample
Enrollment: 250736 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-09-11 (Actual)

PRIMARY OUTCOMES:
Reduction in IL-1β Levels Due to ACE Inhibitors | Baseline to 12 months
  The primary outcome is the reduction in plasma levels of IL-1β due to exposure to ACE inhibitors (ACEIs). The study evaluates the causal relationship between ACEIs and IL-1β levels using Mendelian randomization.（Unit: pg/mL）
Reduction in TNF-α Levels Due to ACE Inhibitors | Baseline to 12 months
  The primary outcome is the reduction in plasma levels of TNF-α due to exposure to ACE inhibitors (ACEIs). The study evaluates the causal relationship between ACEIs and TNF-α levels using Mendelian randomization.（Unit: pg/mL）
Reduction in CRP Levels Due to ACE Inhibitors | Baseline to 12 months
  The primary outcome is the reduction in plasma levels of CRP due to exposure to ACE inhibitors (ACEIs). The study evaluates the causal relationship between ACEIs and CRP levels using Mendelian randomization.（Unit: mg/L）
Modulation of MCP-1 Levels Due to Statin Therapy | Baseline to 12 months
  The primary outcome is the modulation of plasma levels of MCP-1 in patients treated with statins (HMG-CoA reductase inhibitors). The study investigates the effect of statins on MCP-1 levels.（Unit: pg/mL）
Modulation of MIP-1α Levels Due to Statin Therapy | Baseline to 12 months
  The primary outcome is the modulation of plasma levels of MIP-1α in patients treated with statins (HMG-CoA reductase inhibitors).（Unit: pg/mL）
Modulation of MIP-1β Levels Due to Statin Therapy | Baseline to 12 months
  The primary outcome is the modulation of plasma levels of MIP-1β in patients treated with statins (HMG-CoA reductase inhibitors).（Unit: pg/mL）
Reduction in IL-1β Levels Due to PCSK9 Inhibitors | Baseline to 12 months
  The primary outcome is the reduction in plasma levels of IL-1β in individuals exposed to PCSK9 inhibitors.（Unit: pg/mL）
Reduction in IL-6 Levels Due to PCSK9 Inhibitors | Baseline to 12 months
  The primary outcome is the reduction in plasma levels of IL-6 in individuals exposed to PCSK9 inhibitors.（Unit: pg/m）

SECONDARY OUTCOMES:
Reduction in Cardiovascular Events Due to Antihypertensive Therapy | Baseline to 24 months
  The secondary outcome evaluates the reduction in cardiovascular events (e.g., myocardial infarction, stroke) linked to antihypertensive therapies such as ACEIs and ARBs.
Changes in LDL-C Levels Due to Statin Therapy | Baseline to 24 months
  This outcome examines changes in LDL cholesterol (LDL-C) levels due to statin therapy.
Changes in HDL-C Levels Due to Statin Therapy | Baseline to 24 months
  This outcome examines changes in HDL cholesterol (HDL-C) levels due to statin therapy.
Reduction in IL-1β Levels Due to PCSK9 Inhibitors | Baseline to 24 months
  The secondary outcome measures the reduction in IL-1β levels linked to PCSK9 inhibitors.
Changes in Cardiometabolic Outcomes Due to PCSK9 Inhibitors | Baseline to 24 months
  This secondary outcome measures changes in cardiometabolic outcomes, including changes in lipid levels and inflammatory cytokine profiles.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Institute of Respiratory Diseases, the First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) including de-identified genome-wide association study (GWAS) data and inflammatory cytokine levels will be shared. The data will be made available to qualified researchers upon request, following appropriate approval.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available starting 6 months after publication and will be accessible for a period of 5 years.
Access Criteria: Researchers requesting access to the data will need to submit a detailed study proposal and obtain approval from the study's governing ethics board.

REFERENCES:
- [Derived] Xin J, Xu Z, Zhang F, Sun Y, Wang X, Wu C, Zhao L. Mendelian randomization-based observational cohort study on drug targets: Impact of antihypertensive and lipid-lowering therapies on inflammatory cytokines. Medicine (Baltimore). 2025 Mar 7;104(10):e41771. doi: 10.1097/MD.0000000000041771. PMID 40068040